CLINICAL TRIAL: NCT07303049
Title: Cognitive Benefit of Intensive Rehabilitation Using Rhythmic Music Training in Children With Complex Neurodevelopmental Disorder
Acronym: CHUpercu
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/24/0541; ID-RCB : 2025-A01672-47 (Other: ANSM)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Complex Neurodevelopmental Disorder
Keywords: Complex neurodevelopmental disorder; Intensive rhythmic rehabilitation; Cognition; SCED; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with complex neurodevelopmental disorders undergoing intensive rhythmic musical training (Experimental)
  Interventions: Behavioral: Intensive rhythmic musical training

INTERVENTIONS:
Behavioral: Intensive rhythmic musical training — Participants undergo an intensive rhythmic training program using percussion instruments. The program takes place over one week, with daily sessions focused on rhythmic exercises. It focuses on developing motor coordination, timing, and cognitive skills through group-based rhythmic exercises and activities. Sessions include guided percussion practice designed to improve sensorimotor integration and enhance cognitive-motor performance.

SUMMARY:
In the wide range of studies carried out on neurodevelopmental disorders (NDD), rhythm disorders have been identified as a major cross-cutting component. The aim of our research is to evaluate the effect of intensive rhythm-based rehabilitation on rhythmic abilities and its generalization to attentional, executive and reading skills.

DETAILED DESCRIPTION:
Current knowledge of impaired rhythmic skills in NDD is based on a number of studies, mainly carried out with groups of children presenting either Attention Deficit Disorder with or without Hyperactivity (ADHD), Developmental Coordination Disorder (DCD) or Learning to Read Disorder (dyslexia, DYS). The authors highlighted an impairment of the temporal sphere, and more specifically a timing deficit. A few studies have already evaluated the effect of rhythm-based rehabilitation in children with isolated NDD (Flaugnacco et al., 2015; Habib et al., 2013; Jamey et al., 2024; Puyjarinet et al., 2020) and show an improvement in certain untrained cognitive functions (reading skills, phonological awareness, attention, working memory, inhibition).

The intervention, in groups of 6 children, takes place face-to-face, during a school vacation period over 5 consecutive days, 4 hours per day. The sessions are based on specific multimodal training and motor response using the djembe.

After an inclusion visit, all patients undergo a full neuropsychological assessment, which is repeated 2 months later (before-after design). These measurements will take place over one day at the Toulouse University Hospital, in person.

In the meantime, measurements of the assessment criteria are repeated daily before, during and after the intervention, according to a Single Case Experimental Design (SCED). Daily assessments, excluding weekends, will be performed and recorded via the Toulouse University Hospital's TéléO tool. A 5-days final evaluation phase will be carried out 3 months after the intervention to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neurodevelopmental disorder involving at least two impairments (ADHD + DCD, ADHD + Dyslexia, Dyslexia + DCD, ADHD + Dyslexia + DCD), according to DSM-5 criteria (2015), established at the Language and Learning Disorders Reference Center (CRTLA) of Toulouse University Hospital.
* Aged between 8 years and 10 years 6 months.
* Enrolled in elementary school.
* Visual, auditory (with permitted aids), motor, oral and written expression and comprehension abilities sufficient, according to the investigator physician's assessment, to perform cognitive tests and follow the intervention.
* Patient beneficiary/affiliate of the French Social Security system.
* Signed informed consent from parent(s) / legal guardian(s) in accordance with French law and Good Clinical Practice, along with minor's assent.
* Authorization for image and sound recording.

Exclusion Criteria:

* Practice of a musical instrument during the current year (in a music school or leisure activity).
* Behavioral disorder making group practice difficult (e.g., oppositional defiant disorder) according to the investigator's opinion.
* Patient diagnosed with autism spectrum disorder or intellectual developmental disorder (IQ < 70).
* Patient with epilepsy (with or without treatment).
* Uncorrected hearing or visual impairment.
* Current treatment with psychostimulants or psychotropic drugs (notably methylphenidate, antidepressants).
* Patient lacking access to a stable internet connection required for teleconsultation assessments.
* Any family or sociological condition preventing compliance with the procedures outlined in the study protocol, according to the investigator's opinion.
* Patient participating in another human research study involving experimental treatment or behavioral therapy.
* Ongoing rehabilitative care is not an exclusion criterion for the study.

Ages: 8 Years to 126 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rhythmic structure reproduction task (Stambak-type test) | From week 2 after enrollment to week 14

SECONDARY OUTCOMES:
Spontaneous tempo tapping task (SCED methodology) | From week 2 after enrollment to week 14
Behavioral observation grid in ecological settings (SCED methodology) | From week 2 after enrollment to week 14
Text reading task (speed/accuracy ratio) (SCED methodology) | From week 2 after enrollment to week 14
Line orientation judgment task (SCED methodology) | From week 2 after enrollment to week 14
Explicit sensorimotor timing: Synchronization tapping task with a metronome | Week 1 and week 17
Explicit perceptual timing: Beat alignment task | Week 1 and 17
Implicit motor timing (emergent timing): DALS (Draw A Line Slowly) | Week 1 and week 17
Implicit motor timing (emergent timing): WALS (Walk A Line Slowly) | Week 1 and week 17
Selective visual attention: Barre-Joe Test | Week 1 and week 17
Auditory attention: Auditory attention and associated response test | Week 1 and week 17
Planning: 8 Maze Test or Rey-Osterrieth Complex Figure with planning instructions | Week 1 and week 17
Cognitive flexibility: Children's Card Sorting Test - KCST | Week 1 and week 17
Inhibition: Child Tapping Test | Week 1 and week 17
Auditory-verbal: Digit Span Task | Week 1 and week 17
Visuospatial: Spatial memory task | Week 1 and week 17
Pseudoword reading: Evaléo (ages 6-15) | Week 1 and week 17
Text reading: Evaléo (ages 6-15), Forms A and B | Week 1 and week 17
Test assessing passive lexical knowledge: Evaléo (ages 6-15) | Week 1 and week 17
Rapid color naming task: Evaléo (ages 6-15) | Week 1 and week 17
Tapping subtest from NEPSY-II | Week 1 and week 17
Manual dexterity (MABC-2) | Week 1 and week 17
Temporal questionnaire for children (QTE) | Week 1 and week 17
MDI-C (Children's Depression Inventory: Self-esteem subscale, ages 8-17) | Week 1 and week 17
Parent questionnaire: Strengths and Difficulties Questionnaire (SDQ-Fra) | Week 1 and week 17
Child self-assessment from a predefined list of daily activities that may pose difficulties (ecological assessment) | Week 1 and week 17
Likert scale assessing satisfaction across various criteria | Week 17 after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Purpan, Toulouse, Occitanie, France